CLINICAL TRIAL: NCT01291199
Title: Double-blind, Placebo-controlled Cross-over Study to Investigate the Effects of the Phosphodiesterase 5-inhibitor Vardenafil on Periphery Blood Flow and Clinical Symptoms of Patients With Raynaud's Syndrome
Brief Title: Effects of Vardenafil on Clinical Symptoms and Peripheral Blood Flow in Patients With Raynaud's Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Prof. Dr. med. Erland Erdmann, Universität zu Köln
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ro-002/05; 2005-000295-41 (EudraCT Number)
Record Dates: First submitted 2011-02-01; First posted 2011-02-08 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-01

CONDITIONS: Raynaud Syndrome
Keywords: double-blind placebo controlled cross-over study
MeSH Terms: conditions — Raynaud Disease | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vardenafil 10 mg bid (Experimental)
  Interventions: Drug: vardenafil; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: vardenafil; Drug: Placebo

INTERVENTIONS:
Drug: vardenafil — 10 mg p.o. bid for 6 weeks
  Other Names: Levitra
Drug: Placebo — Placebo p.o. 6 weeks bid

SUMMARY:
The purpose of this study is to determine whether vardenafil is effective in improving clinical symptoms and peripheral blood flow in patients with primary and secondary Raynaud phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* raynaud-syndrome (primary or secondary) > 1 year duration
* age ≥ 18 years; ≤ 80 years
* informed consent
* a negative pregnancy test in women of child-bearing age

Exclusion Criteria:

* any unstable organic, psychiatric or addictive disease, which - in the opinion of the investigators - might result in an unsuccessful / unreliable participation or premature termination of the trial
* known contraindications against PDE 5-inhibitors (such as intolerance, therapy with nitrates or inhibitors of CYP3A4, etc.)
* extensive necrosis of the finger tips
* pigmentary retinopathy
* verification as a HbsAg or hepatitis C carrier
* unstable angina
* heart failure (NYHA III or IV)
* valve defects of higher degree (particularly aortic stenosis and hypertrophic obstructive cardiomyopathy)
* myocardial infarction, stroke or life-threatening cardiac arrhythmias within the last 6 months
* uncontrolled atrial fibrillation / -flutter with a heart rate > 100 bpm
* prolonged QTc-interval (> 450 msec)
* congenital long-QT-syndrome
* hypokalemia
* severe acute or chronic liver disease, which might lead to priapism (sickle cell anemia, leucemia)
* hemophilia
* active peptic ulcers
* arterial hypotension (systolic blood pressure at rest <90 mmHg) or
* arterial hypertension(systolic blood pressure at rest >170 mmHg or diastolic blood pressure at rest >110 mmHg)
* malignancy within the last 5 years (except squamous or basal cell skin cancer)
* patients with injuries of the spinal cord or central nervous system
* patients with severe chronic kidney disease (creatinin clearance < 30 ml)
* patients with mild to severe liver disease (Child-Pugh A-C)
* Age below 18 or above 80
* prohibited concomitant medication during the study:

  * nitrates or other NO-donators (including amylnitrit)
  * anticoagulative drugs except inhibitors of thrombocyte function
  * androgens (such as testosterone) or anti-androgens
  * strong inhibitors of cytochrome P4503A4:
* very potent HIV-Protease-inhibitors (ritonavir, indinavir)
* anti-mycotic like itraconazole and ketoconazole (topical applications are allowed)
* erythromycin
* grapefruit-juice or products containing grapefruit-juice

  * other study medications (including placebo) up to 30 days before study inclusion
  * therapy of erectile dysfunction(including sildenafil, sublingual apomorphin, MUSE®, intracavernous injections or vacuum pumps) or other therapies of erectile dysfunction within 4 weeks and during the trial period
  * nebivolol
  * alpha-blockers
  * Calcium antagonists
  * medications prolonging the QT-interval
  * abnormal lab tests like:
* serum-creatinine > 3 mg/dl at visit 1
* GOT and GPT > 3 x reference limit set
* diabetes mellitus with a HbA1c > 9%
* patients who are not willing to disclaim a therapy of their erectile dysfunction with vacuum pumps, intravenous injections, sildenafil or other therapies during the trial
* severe migraine (more than once a moth during the last 6 months)
* intolerance to the study medication
* patients who are not able to understand the information and informed consent due to a mental disorder or linguistic barriers
* persons who are living in a institution directly under federal government control due to a court order
* patients who refuse to renounce drinking grapefruit juice during the trial
* women who are pregnant or lactating
* women who are not protected from a pregnancy (intake of oral contraceptives alone in insufficient; highly effective methods of birth control have to be used with a failure rate <1%; barriers: implants, intrauterine-devices (IUD´s),diaphragm, condoms, abstinence, partner is vasectomized, spermicides)
* patients who participated in other interventional studies within 30 days of study inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-11; Primary Completion 2009-08 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in the Raynaud's Condition Score | daily for 18 weeks
  The Raynaud's Condition Score (RCS) is a clinically validated scale used to determine the difficulty that patients experience with Raynaud's phenomenon, and is closely associated with the measures of disability and overall impact and activity of the disease.

SECONDARY OUTCOMES:
Number of participants with adverse events as a Measure of Safety and Tolerability | daily for 18 weeks
Digital blood flow | at baseline, one hour after drug intake and after six weeks on therapy
  digital blood flow measured with laser doppler

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Rosenkranz, MD, Principal Investigator — University of Cologne
Locations (1):
- University of Cologne - Heart Center, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Caglayan E, Huntgeburth M, Karasch T, Weihrauch J, Hunzelmann N, Krieg T, Erdmann E, Rosenkranz S. Phosphodiesterase type 5 inhibition is a novel therapeutic option in Raynaud disease. Arch Intern Med. 2006 Jan 23;166(2):231-3. doi: 10.1001/archinte.166.2.231. PMID 16432094